CLINICAL TRIAL: NCT06371105
Title: Effect of Water-based Aerobic Training on Anthropometric, Biochemical, Cardiovascular, and Explosive Strength Parameters in Young Overweight and Obese Women
Brief Title: Aquatic_Training in Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Taipei (Other)
Responsible Party: Principal Investigator, YUNG-SHENG CHEN, Professor, University of Taipei
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 014_2018
Record Dates: First submitted 2024-03-28; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Obesity
Keywords: aquatic training; body composition; lipid profile; obesity management; physical fitness testing; resting heart rate
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): Performing a 10-week water-based aerobic training (thrice/week)
  Interventions: Other: 10-week water-based aerobic training
- Control group (No Intervention): Maintaining their usual activities during the interventional period

INTERVENTIONS:
Other: 10-week water-based aerobic training — The water-based aerobic program was adopted from the protocol previously used by Costa et al. (2018, 2020). This training program was carried out thrice a week over 2 non-consecutive days 48 hours apart for 10 weeks according to ACSM guidelines
  Arms: Training group

SUMMARY:
This study aims to assess the effects of 10-week water-based aerobic training (thrice a week) on anthropometrics, biochemicals, cardiovascular parameters, and explosive strength in young overweight and obese women. The findings indicate that water-based aerobic training could be a useful program to enhance body composition, biochemical, cardiovascular, and explosive strength parameters in young overweight and obese women compared to inactive persons

DETAILED DESCRIPTION:
This study is based on a randomized controlled trial with a pre-to-post testing design, twenty-seven young overweight and obese women were assigned to training group (a water-based aerobic training) or control group (maintaining their usual activities during the studying period. For each training session, water activities were implemented for 50 min which included warm-up (10 min), main activities (30 min), and cool-down (10 min). The swimming pool where the intervention took part was 1.50 m deep of water. The pre- and post-intervention participants were assessed for their anthropometrics, biochemicals (fasting glycemia, total cholesterol, high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol and triglyceride (TG)), resting blood pressure, and resting heart rate, and explosive strength of upper (countermovement jump and squat jump) and lower limbs (a seated medicine ball throw test).

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 35 years
* Sedentary lifestyle within six month
* Not using drugs or other therapy for obesity.

Exclusion Criteria:

* BMI below 25.0 and over 34.9 kg.m-2
* having any infectious or skin diseases

Ages: 29 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
fasting glycemia in millimoles per liter | 3 days before the 10-week interventional period
  baseline blood sample
total cholesterol in millimoles per liter | 3 days before the 10-week interventional period
  baseline blood sample
high-density lipoprotein cholesterol in millimoles per liter | 3 days before the 10-week interventional period
  baseline blood samplelipoprotein cholesterol, and triglyceride concentrations
low-density lipoprotein cholesterol in millimoles per liter | 3 days before the 10-week interventional period
  baseline blood sample
triglyceride concentrations in millimoles per liter | 3 days before the 10-week interventional period
  baseline blood sample
systolic blood pressure in millimeters of mercury | 3 days before the 10-week interventional period
  baseline blood sample
diastolic blood pressure in millimeters of mercury | 3 days before the 10-week interventional period
  baseline blood sample
heart rate in beat per minute | 3 days before the 10-week interventional period
  baseline blood sample
fasting glycemia in millimoles per liter | one day after the 10-week interventional period
  post-training blood sample
total cholesterol in millimoles per liter | one day after the 10-week interventional period
  post-training blood sample
high-density lipoprotein cholesterol in millimoles per liter | one day after the 10-week interventional period
  post-training blood sample
low-density lipoprotein cholesterol in millimoles per liter | one day after the 10-week interventional period
  post-training blood sample
triglyceride concentrations in millimoles per liter | one day after the 10-week interventional period
  post-training blood sample
systolic blood pressure in millimeters of mercury | one day after the 10-week interventional period
  post-training blood sample
diastolic blood pressure in millimeters of mercury | one day after the 10-week interventional period
  post-training blood sample
heart rate in beat per minute | one day after the 10-week interventional period
  post-training blood sample

SECONDARY OUTCOMES:
countermovement jump in centimetres | 3 days before the 10-week interventional period
  baseline lower limbs power test
squat jump in centimeters | 3 days before the 10-week interventional period
  baseline lower limbs power test
chest 3-kg medicine ball throw in meters | 3 days before the 10-week interventional period
  baseline upper limbs power test
countermovement jump in centimetres | one day after the 10-week interventional period
  post-training lower limbs power test
squat jump in centimeters | one day after the 10-week interventional period
  post-training lower limbs power test
chest 3-kg medicine ball throw in meters | one day after the 10-week interventional period
  post-training upper limbs power test

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Sheng Chen, Ph.D., Study Director — Department of Exercise and Health Sciences, University of Taipei
Locations (1):
- Department of Exercise and Health Sciences, University of Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No